CLINICAL TRIAL: NCT06683326
Title: Smart-gloves Hand Motion Tracking for Live Endoscopic Submucosal Dissection Training: a Randomized, Comparative Study
Brief Title: Smart-gloves Hand Motion Tracking for Live Endoscopic Submucosal Dissection Training
Acronym: EndoHandView
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Mihai Ciocirlan, Associate Professor, Carol Davila University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EndoHandView
Record Dates: First submitted 2024-10-28; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Animal Model
MeSH Terms: conditions — Disease Models, Animal

STUDY DESIGN:
Intervention Model Description: Two randomized groups of trainees.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Trainees viewing live broadcasting of the ESD screen, with live explanations by the expert and simultaneous viewing of the expert hands and fingers motion broadcasted by the ROKOKO smart-glove.
  Interventions: Device: ROKOKO smart-glove
- Control group (No Intervention): Control group, trainees viewing live broadcasting of the ESD screen, with live explanations by the expert

INTERVENTIONS:
Device: ROKOKO smart-glove — ESD expert hands and fingers motion broadcasted by the ROKOKO smart-glove to trainees
  Arms: Study group

SUMMARY:
Learning endoscopic submucosal dissection (ESD) is undertaken by experienced endoscopists in endoscopic mucosal resection and management of complications. Understanding the theoretical approach of the procedure and the cutting line is a prerequisite of performing it. The precise knife movements following the cutting line during incision, trimming and dissection takes time to master.

The European Society of Gastrointestinal Endoscopy (ESGE) recommends certain steps of the learning process: starting on animal models and further passing onto easier cases in patients, all these with expert supervision. Observation of experts directly or in live endoscopy meetings are recommended. Direct observation of the experts allow viewing and understanding the hand and finger movements during the specific ESD procedure phases (incision, trimming, dissection). Conversely, during live endoscopy meetings, one cannot see the hand and fingers movements of the operator. Using motion tracking smart-gloves, these fine movements may be visually broadcasted together with the endoscopic view during live meetings. There currently are no studies on motion tracking of hand and finger movements smart gloves in gastrointestinal endoscopy.

Broadcasting the ESD expert's hands and fingers movements using a motion tracking smart-glove during a live endoscopy event will increase the trainees ESD procedure speed. Concomitantly seeing the endoscopic view and the hand and fingers view, the trainee will establish a relationship between the hand and fingers movement and the effect on the dissected tissue. A faster practical "how to do it" formula will hopefully be acquired by the trainee.

Additional benefits are expected, as a faster trainee learning curve will diminish the carbon footprint of the endoscopic training process.

A prospective randomized study will be implemented to test the research hypothesis. Trainees will be divided in two groups, depending on their view during live ESD procedures performed by the experts: the study group [endoscopic view + hand motion view] versus the control group [only endoscopic view]. The experts endoscopists will demonstrate ESD procedures on an animal model. Afterwards, the trainee will perform, under supervision, an ESD procedure on the same animal model. Several parameters will be noted: speed of the procedure, the en-bloc or piece-meal resection, the R0 resection, presence of complications (perforation) and the satisfaction score of the trainee on a numerical visual scale.

DETAILED DESCRIPTION:
Rationale.

ESD is difficult to learn. Learning is usually undertaken by already trained endoscopists, with experience in difficult polypectomy. Except marking, hemostasis and clip closure, the very precise distinctive ESD movements - incision, trimming and submucosal dissection are new hand gestures for someone starting this path.

After studying ESD strategy and tactics - where to start and continue ("when to cut") and what part of the lesion ("what to cut"), one needs to understand the cutting line ("where to cut"). This cutting line is to be followed precisely, in an extremely accurate manner during incision, trimming and actual submucosal dissection. Any millimetric deviation from this ideal line may and will result in lengthening or procedure failure in best case scenario and in iterative bleedings and perforation in worst case scenarios.

The ESGE learning curricula recommends that a proficient in EMR endoscopist should start supervised ESD training. Firstly, in animal models (at least 20 procedures with no perforation in the last 10 training cases and 80% R0 rate) and afterwards, supervised simpler cases on real patients [1]. Observing at least 20 ESD procedures performed by experts in tertiary referral centers as well as live conferences and meetings are encouraged.

Based on available evidence, current ESGE and ASGE guidelines for best practices of live endoscopy events do not find an increased harm for patients [2,3]. Moreover, in a study comparing the outcomes of ESD in a live event versus standard of care, the outcome numbers were non-inferior, and some were even slightly non significantly superior (en-bloc rates 100% vs. 87%, curative rates 84% vs. 71%, complication rates 5% vs. 13%, 5-year survival rates 70% vs. 65%) [4]. Nevertheless, both guidelines state that there is no current data supporting that attending live endoscopy events will improve ESD outcome in trainees.

Unfortunately, observing an ESD procedure during a live endoscopy event is not the same experience as being in the same room as the operator. The endoscopic screen and the verbal explanations may be there. Still, the exact hand movements by the operator will be missed. Viewing the expert's hands and fingers movements during such a complex procedure is of utmost importance.

A recent 2023 study evaluated the benefit of a live broadcasting GoPro action camera attached to the endoscopist head [5]. The supplementary doctor's eye-view video increased the trainees interest and understanding of the procedure. However, as the endoscopist gaze will be pointed to the endoscopy screen most of the time, the hand and finger gestures will not be GoPro broadcasted and live seen by trainees.

How to observe and analyze hand and finger movements during and ESD procedure? Hand gestures during colonoscopy were quantified in different studies assessing pressure and force by tactile pads, electrogoniometers, magnetic trackers and electromagnetic motion sensors [6-9]. These studies aimed to assess muscle strain and postures during colonoscopy and their different patterns in expert and novice operators.

Smart-gloves were proposed to measure kinesthetic and tactile feed-back, but also hand and finger pose and motion tracking [10]. Medical studies so far used hand motion tracking smart-gloves to quantify and/or monitor concomitant brain activation, hand joints stress, chest compressions during CPR, drawing coordination skills, surgical knot tying and post stroke hand grip rehabilitation [11-16]. Tracking hand and fingers motion during ESD may be possible as well using available commercial smart-gloves.

The ROKOKO smart-gloves use electro-magnetic field (EMF) sensors to capture precise hand and finger movements. It instantly broadcasts with 100 frame per second rate, without lag or latency. It may be integrated with all major 3D animation tools and game engines and is currently used, among others, by Walt Disney Studios, Universal Studios, Sony, Netflix, HBO, Electronic Arts, [17].

Study hypothesis.

Broadcasting the ESD expert's hands and fingers movements using a motion tracking smart-glove during a live endoscopy event will increase the trainees speed of the ESD procedure. It will increase the rate of en-bloc resection, the rates of curative resection and will decrease the rate of complications. While at distance, the trainee will be able to concomitantly see the two screens - the [endoscopic view] and the [hand and fingers view]. A relationship between the hand and fingers motions and the transmitted effect onto knife tip and further onto the lesion tissue will be better understood. A practical "how to do it" knowledge will be hopefully acquired by the trainee, faster.

ELIGIBILITY:
Inclusion Criteria:

* ESD trainees with experience in EMR and difficult polypectomy

Exclusion Criteria:

* ESD trainees with previous significant experience in ESD on animal model
* ESD trainees with previous significant experience in ESD on patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Mean speed of the procedure | During procedure
  Measured in mm2/minute. Equal to the sum of the procedure speed for each procedure divided by the number of procedures for each study group.

SECONDARY OUTCOMES:
Rate of en-bloc resection | During procedure
  Defined as lesions resected in one piece. Equal to the number of en-bloc resected lesions divided by the number of resected lesions for each study group.
Rate of R0 resection. | During procedure
  Defined as lesions resected in one piece containing all peripheral marking dots. Equal to the number of R0 resections divided by the number of resected lesions in each group.
Rate of perforation. | During procedure
  Equal to the number of perforations divided by the number of resected lesions in each group.
Median satisfaction score. | Immediately after procedure
  Measured on a visual analogue scale (0 to 10, 0 equal unsatisfied, 10 equal maximum satisfaction). Equal to the median satisfaction value of trainees within each study group.

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Ciocirlan, MD, Principal Investigator — Carol Davila University of Medicine and Pharmacy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pimentel-Nunes P, Pioche M, Albeniz E, Berr F, Deprez P, Ebigbo A, Dewint P, Haji A, Panarese A, Weusten BLAM, Dekker E, East JE, Sanders DS, Johnson G, Arvanitakis M, Ponchon T, Dinis-Ribeiro M, Bisschops R. Curriculum for endoscopic submucosal dissection training in Europe: European Society of Gastrointestinal Endoscopy (ESGE) Position Statement. Endoscopy. 2019 Oct;51(10):980-992. doi: 10.1055/a-0996-0912. Epub 2019 Aug 30. PMID 31470448
- [Background] Webster GJ, El Menabawey T, Arvanitakis M, Hassan C, van Hooft JE, Messmann H, Dinis-Ribeiro M. Live endoscopy events (LEEs): European Society of Gastrointestinal Endoscopy Position Statement - Update 2021. Endoscopy. 2021 Aug;53(8):842-849. doi: 10.1055/a-1511-1657. Epub 2021 Jun 10. PMID 34111899
- [Background] Khashab MA, Muthusamy VR, Akshintala VS, Kothari S, Sethi A, Rastogi A, Palmisano DJ Jr, Zhang LY, Hess MR, Rashba K, Gupta N, Wani S, Komanduri S. Best live endoscopy practices: an ASGE white paper. Gastrointest Endosc. 2023 Mar;97(3):383-393.e3. doi: 10.1016/j.gie.2022.09.012. Epub 2023 Jan 11. No abstract available. PMID 36639318
- [Background] Ebigbo A, Freund S, Probst A, Rommele C, Golder SK, Frauenschuh J, Marienhagen J, Messmann H. Outcomes of endoscopic submucosal dissection (ESD) during live endoscopy events (LEE) - a 13-year follow-up. Endosc Int Open. 2019 Dec;7(12):E1723-E1728. doi: 10.1055/a-1035-9240. Epub 2019 Dec 10. PMID 31828208
- [Background] Uchiyama A, Yamashina S, Sato T, Sakuma S, Tomiki Y, Isayama H, Nagahara A, Ikejima K. Benefit of an action camera in endoscopy education for medical students under COVID-19. BMC Med Educ. 2023 Sep 22;23(1):693. doi: 10.1186/s12909-023-04702-6. PMID 37740173
- [Background] Shergill AK, Asundi KR, Barr A, Shah JN, Ryan JC, McQuaid KR, Rempel D. Pinch force and forearm-muscle load during routine colonoscopy: a pilot study. Gastrointest Endosc. 2009 Jan;69(1):142-6. doi: 10.1016/j.gie.2008.09.030. PMID 19111694
- [Background] Browne A, O'Sullivan L. A medical hand tool physical interaction evaluation approach for prototype testing using patient care simulators. Appl Ergon. 2012 May;43(3):493-500. doi: 10.1016/j.apergo.2011.08.002. Epub 2011 Aug 30. PMID 21880299
- [Background] Mohankumar D, Garner H, Ruff K, Ramirez FC, Fleischer D, Wu Q, Santello M. Characterization of right wrist posture during simulated colonoscopy: an application of kinematic analysis to the study of endoscopic maneuvers. Gastrointest Endosc. 2014 Mar;79(3):480-9. doi: 10.1016/j.gie.2013.11.023. Epub 2014 Jan 17. PMID 24439784
- [Background] Holden MS, Wang CN, MacNeil K, Church B, Hookey L, Fichtinger G, Ungi T. Objective assessment of colonoscope manipulation skills in colonoscopy training. Int J Comput Assist Radiol Surg. 2018 Jan;13(1):105-114. doi: 10.1007/s11548-017-1676-4. Epub 2017 Oct 30. PMID 29086234
- [Background] Caeiro-Rodriguez M, Otero-Gonzalez I, Mikic-Fonte FA, Llamas-Nistal M. A Systematic Review of Commercial Smart Gloves: Current Status and Applications. Sensors (Basel). 2021 Apr 10;21(8):2667. doi: 10.3390/s21082667. PMID 33920101
- [Background] Brand J, Piccirelli M, Hepp-Reymond MC, Eng K, Michels L. Brain Activation During Visually Guided Finger Movements. Front Hum Neurosci. 2020 Aug 14;14:309. doi: 10.3389/fnhum.2020.00309. eCollection 2020. PMID 32922274
- [Background] Jaskiewicz F, Kowalewski D, Starosta K, Cierniak M, Timler D. Chest compressions quality during sudden cardiac arrest scenario performed in virtual reality: A crossover study in a training environment. Medicine (Baltimore). 2020 Nov 25;99(48):e23374. doi: 10.1097/MD.0000000000023374. PMID 33235109
- [Background] Lee HS, Lim JH, Jeon BH, Song CS. Non-immersive Virtual Reality Rehabilitation Applied to a Task-oriented Approach for Stroke Patients: A Randomized Controlled Trial. Restor Neurol Neurosci. 2020;38(2):165-172. doi: 10.3233/RNN-190975. PMID 32176674
- [Background] Lacroute J, Marcantoni J, Petitot S, Weber J, Levy P, Dirrenberger B, Tchoumak I, Baron M, Gibert S, Marguerite S, Huppertz J, Gronier O, Derlon A. The carbon footprint of ambulatory gastrointestinal endoscopy. Endoscopy. 2023 Oct;55(10):918-926. doi: 10.1055/a-2088-4062. Epub 2023 May 8. PMID 37156511
- See also: Lacey G, Ridgway P, Bhattacharya J. Measuring surgical knot tying with 3D vision and VR gloves. Semantic Scholar. 2019; — https://www.semanticscholar.org/paper/Measuring-surgical-knot-tying-with-3D-vision-and-VR-Lacey-Ridgway/012bf54cc7728bd4cf96bb0892e6e4e1c32f9bb9
- See also: https://www.rokoko.com/ — https://www.rokoko.com/
- See also: https://www.randomizer.org — https://www.randomizer.org